CLINICAL TRIAL: NCT04310540
Title: Development and Validation of Innovative Hybrid Molecular Imaging, 68Ga-PSMA-Dual Contrast PET/MRI and 68Ga-PSMA PET/CT, to Transform the Care of Patients with Hepatocellular Carcinoma
Brief Title: PSMA PET/MRI or PSMA PET/CT for Evaluation of Liver Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-012563; NCI-2021-02760 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Biopsy; gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (gallium Ga 68 gozetotide PET/MRI, PET/CT, biopsy) (Experimental): Patients receive gallium Ga 68 gozetotide IV, and undergo PET/MRI over 60 minutes or PET/CT over 30 minutes at baseline and 12 weeks after completion of hepatic locoregional therapy or 8-12 weeks after completion of systemic therapy. Patients undergoing hepatic locoregional therapy may also undergo a liver biopsy.
  Interventions: Procedure: Biopsy; Procedure: Computed Tomography; Drug: Gallium Ga 68 Gozetotide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This clinical trial evaluates whether 68Ga-PSMA PET/MRI or PET/CT can improve upon the diagnosis and management of liver cancer. MRI stands for magnetic resonance imaging, a scan that uses magnetic and radio waves to produce detailed structural information of the organs, tissues and structures within the body. PET stands for positron emission tomography, an imaging test that helps to measure the information about functions of tissues and organs within the body. A PET scan uses a radioactive drug (radiotracer) to show this activity. CT scan uses X-rays to create images of the bones and internal organs within the body. In patients that have been diagnosed with liver cancer, a protein called prostate specific membrane antigen (PSMA) appears in large amounts on the surface of the cancerous cells. The radioactive chemical compound (68Ga-PSMA) has been designed to circulate through the body and attach itself to the PSMA protein on liver cancer cells. 68Ga-PSMA PET/MRI or PET/CT may be better in diagnosing and managing liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate diagnostic performance of gallium Ga 68 gozetotide (68Ga-PSMA-dual contrast [Gadavist and gadoxetate]) positron emission tomography (PET)/magnetic resonance imaging (MRI) OR PET/computed tomography (CT) for hepatocellular carcinoma (HCC) using surgical histopathology (either resection, transplant or biopsy specimens) or Liver Imaging and Reporting Data System (LI-RADS) categorization as gold standard.

II. To evaluate treatment response after locoregional therapy or systemic therapy in HCC using 68Ga-PSMA uptake at PET (qualitative & semi-quantitative measures) and to compare it with standard CT/MRI morphologic and post-contrast enhancement based response criteria (modified Response Evaluation Criteria in Solid Tumors [mRECIST] and LI-RADS-treatment response [LR-TR] algorithm).

III. To determine association between PSMA uptake in HCCs at PET with tissue prostate specific membrane antigen (PSMA) expression using immunohistochemistry or serum/plasma PSMA expression using enzyme-linked immunosorbent assay (ELISA).

OUTLINE:

Patients receive gallium Ga 68 gozetotide intravenously (IV), and undergo PET/MRI over 60 minutes or PET/CT over 30 minutes at baseline and 12 weeks after completion of hepatic locoregional therapy or 8-12 weeks after completion of systemic therapy. Patients undergoing hepatic locoregional therapy may also undergo a liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either an imaging diagnosis of HCC by CT or MRI (LI-RADS 5) confirmed by a board-certified abdominal radiologist, or with biopsy-proven HCC
* Subjects who may undergo hepatic surgical resection, liver transplant, hepatic locoregional therapy (ablation, embolization, etc.) or systemic therapy
* No prior treatment for index HCC lesion (surgical resection, liver transplant, hepatic locoregional therapy arm)
* For the systemic therapy arm, patients who have had unequivocal progression after prior locoregional therapy (LRT) and/or those undergoing de novo systemic therapy in view of advanced HCC at diagnosis
* Male or female with age greater than 18 years, with the capacity and willingness to provide a written informed consent

Exclusion Criteria:

* Subjects requiring emergent surgery for a ruptured/bleeding HCC
* Bilirubin > 3.0 mg/dL, which is a contraindication for Gadoxetate, the MRI contrast agent (relevant to PET/MRI)
* Pregnant and/or breast-feeding subjects. A negative pregnancy test within 48 hours of the PET scan
* Subjects with higher than the weight/size limitations of PET/MRI or PET/CT scanner
* Subjects with contraindication to MRI (relevant to PET/MRI):

  * Subjects who have a heart pacemaker
  * Subjects who have a metallic foreign body (metal sliver) in their eye, or who have an aneurysm clip in their brain
  * Subjects who have implanted devices with magnets
  * Subjects who have other implanted electronic devices
  * Subjects who have deep brain stimulator
  * Subjects who have vagal nerve stimulator
  * Subjects with cochlear (ear) or auditory implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-11-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of 68Ga-PSMA-dual contrast (gadavist and gadoxetate) positron emission tomography/magnetic resonance imaging (PET/MRI), or 68Ga-PSMA positron emission tomography/computed tomography (PET/CT) | At 3 months after completion of hepatic locoregional therapy or systemic therapy
  Using surgical histopathology (either resection or transplant specimens) or Liver Imaging and Reporting Data System (LI-RADS[R]) categorization as gold standard.
Treatment response after locoregional therapy in hepatocellular carcinoma (HCC) | Completion of locoregional therapy (up to 3 months)
  Using 68Ga-PSMA uptake at PET (qualitative & semi-quantitative measures) compared with standard CT/MRI morphologic and post-contrast enhancement based response criteria (modified Response Evaluation Criteria in Solid Tumors and LI-RADS-treatment response [LR-TR] algorithm).
Association between prostate specific membrane antigen (PSMA) uptake in hepatocellular carcinoma at PET with tissue PSMA expression | Up to 3 years
  Assessed using immunohistochemistry, serum/plasma PSMA expression using enzyme-linked immunosorbent assay or serum HCC tumor markers.

CONTACTS AND LOCATIONS:
Overall Officials: Ajit H. Goenka, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials